CLINICAL TRIAL: NCT03182179
Title: Efficacy of Ondansetron in the Treatment of Low Anterior Resection Syndrome (LARS): a Multi-centre, Randomized, Double Blind, Placebo-controlled Crossover Study
Brief Title: Efficacy of Ondansetron in LARS Treatment
Acronym: Hodolar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORL-CHIR-001
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- O-P sequence (Experimental): Patients will receive of oral Ondansetron 4mg BD for 28 days followed by 28 days of placebo. It will be one week of washout between the two treatments.
  Interventions: Drug: Ondansetron 4 MG; Drug: Placebo
- P-O sequence (Experimental): Patients will receive oral placebo for 28 days followed by Ondansetron 4mg BD for 28 days. It will be one week of washout between the two treatments.
  Interventions: Drug: Ondansetron 4 MG; Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron 4 MG — Ondansetron is taken orally BD
Drug: Placebo — Placebo is taken orally BD

SUMMARY:
Patients will be randomized (1:1 ratio) to receive either 4 weeks of Ondansetron followed by 4 weeks of placebo (O-P sequence) or 4 weeks of placebo followed by 4 weeks of Ondansetron (P-O sequence). It will be one week of washout between the two treatments.

During the treatment questionnaires will be completed by the patients to evaluate the efficacy of the study treatment and the quality of live.

DETAILED DESCRIPTION:
This is a multi-centre randomized, double-blind, placebo-controlled, cross-over study aimed at testing the efficacy of Ondansetron in the low anterior resection syndrome (LARS) occurring as a consequence of surgery for rectal cancer.

Patients will be randomized (1:1 ratio) to receive either 4 weeks of Ondansetron followed by 4 weeks of placebo (O-P sequence) or 4 weeks of placebo followed by 4 weeks of Ondansetron (P-O sequence). Neither the investigator nor the patient will be aware of the sequence (O-P or P-O) assigned to the patient. One week will elapse between the end of the first treatment and start of the second treatment.

The hypothesis to be tested is that 4 weeks of oral Ondansetron at the dose of 4mg BID induce a variation of the LARS Score at least 7 points (20%) greater than the variation occurring after 4 weeks of placebo.

The sample size calculated for the primary analysis is 38 evaluable patients. Considering an expected attrition rate of about 20%, it is expected to enrol approximately 46 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients willing and able to comply with the study procedures
* Female patients of childbearing potential must agree to use a reliable method of contraception
* Written informed consent Patients who have undergone low anterior resection (LAR) for rectal cancer in the last 2 years provided that at least 4 weeks have elapsed since recanalization and 4 weeks have elapsed since any chemo- and/or radiotherapy
* Presence of functioning anastomosis
* Presence of significant LARS symptoms assessed by LARS Score

Exclusion Criteria:

* Known hypersensitivity or allergy to Ondansetron
* Previous Ondansetron antiemetic therapy completed less than 4 weeks before study entry
* Antitumor chemotherapy or radiotherapy completed less than 4 weeks before study entry
* Congenital long Q-T syndrome
* Ongoing treatment with drugs causing prolongation of the Q-T interval
* Uncorrected hypokalemia or hypomagnesemia
* Women who are pregnant or breast feeding or are willing to become pregnant during the study
* Clinically significant concomitant disease states or anastomotic complications which could impair the ability of the patient to participate in the trial
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Change in LARS score | 10 wks
  The primary outcome is the change in LARS Score assessed before and after Ondansetron and placebo treatment

SECONDARY OUTCOMES:
Vaizey (St. Mark's) score | 10 wks
  Change in Vaizey (St. Mark's) Score assessed before and at the end of Ondansetron and placebo treatment
Irritable Bowel Syndrome-Quality of Life | 10 wks
  Irritable Bowel Syndrome-Quality of Life (IBS-QoL) assessed before and at the end of Ondansetron and placebo treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Christoforidis, Prof., Study Director — Ospedale Regionale di Lugano, Civico e Italiano
Locations (2):
- Switzerland (2):
  - CHUV, Lausanne
  - Ospedale Regionale di Lugano, Civico e Italiano, Lugano

IPD SHARING:
Plan to Share IPD: No